CLINICAL TRIAL: NCT06785948
Title: tDCS Effect on Psychotic Symptoms in Dementia With Lewy Bodies (DLB), and Impacts on Caregiver Burden
Acronym: MCL-tDCS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Association de Recherche Bibliographique pour les Neurosciences (Other)
Collaborators: Centre Hospitalier Princesse Grace (Other); Association des Aidants et Malades à Corps de Lewy (A2MCL) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MCL-tDCS
Record Dates: First submitted 2025-01-09; First posted 2025-01-21 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Lewy Body Dementia; Lewy Body Dementia With Behavioral Disturbance; Burden, Caregiver; Lewy Body Disease; Dementia With Lewy Bodies
Keywords: Transcranial Direct-Current Stimulation (t-DCS); Brain stimulation; Psychotic symptoms; Caregiver burden
MeSH Terms: conditions — Lewy Body Disease; Caregiver Burden

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Active Comparator)
  Interventions: Device: active-tDCS
- Sham tDCS (Sham Comparator)
  Interventions: Device: Sham-tDCS

INTERVENTIONS:
Device: active-tDCS — 2mA stimulation (anode on the left dorsolateral prefrontal cortex, cathode on the right fronto-orbital).
  10 sessions of 20 minutes each, spread over 2 consecutive weeks (5 days with stimulation, 2 days without stimulation, 5 days with stimulation).
  Arms: Active tDCS
Device: Sham-tDCS — No intensity applied (anode on the left dorsolateral prefrontal cortex, cathode on the right fronto-orbital).
  10 sessions of 20 minutes each, spread over 2 consecutive weeks (5 days with stimulation, 2 days without stimulation, 5 days with stimulation).
  Arms: Sham tDCS

SUMMARY:
The goal of this pilot prospective study is to evaluate the effect of tDCS on psychotic-like symptoms in patients with Lewy Body Dementia (LBD). The main questions it aims to answer are:

* What is the effect of tDCS on neuropsychiatric symptoms, especially psychotic-like symptoms?
* What is the impact of tDCS on caregiver burden?

Researchers will compare active tDCS (2mA stimulation, anode on the left dorsolateral prefrontal cortex, cathode on the right fronto-orbital) to Sham tDCS (placebo stimulation, no intensity applied) to see if there is an effect on reducing psychotic-like symptoms and on caregiver burden.

Participants will:

* Undergo a stimulation phase consisting of 10 tDCS sessions of 20 minutes each, spread over 2 consecutive weeks (5 days with stimulation, 2 days without stimulation, 5 days with stimulation).
* perform assessments at T0 (inclusion), T1 (at the end of the stimulation phase), and T2 (follow-up at 8 weeks post stimulation).

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, aged over 60,
* Diagnosed with a neurodegenerative pathology of the DLB type, at a moderate stage, according to the McKeith and al. (2017) criteria
* No change in antiparkinsonian or psychotropic medications, or cholinesterase inhibitors, for a period of one month prior to inclusion,
* Mini Mental State Examination (MMSE) > 15,
* Composite score called "psychotic factor" (corresponding to the sum of the psychotic-type symptoms sub-scores from the NPI [12]) greater than 0,
* Presence of a family caregiver,
* Sufficient written and oral expression in French,
* Written informed consent signed by the patient and his/her family caregiver

Exclusion Criteria:

* History of alcoholism, drug addiction or neurological diseases such as brain trauma, epilepsy, encephalitis, intracranial normal-pressure hydrocephalus, etc. which may lead to cognitive impairment,
* Concomitant major psychiatric illness,
* Significant physical illness or comorbidities
* History of moderate to severe visual impairment secondary to glaucoma, cataract or macular degeneration,
* Patient under guardianship or curators

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the composite score named "psychotic factor" at T1 | Baseline, Week 2
  "psychotic factor" corresponds to the sum of the subscores of psychotic-like symptoms from the Neuropsychiatric Inventory (NPI), namely Delusions, Hallucination, and Agitation/Aggression.
Change from Baseline in the composite score named "psychotic factor" at T2 | Baseline, Week 10
  "psychotic factor" corresponds to the sum of the subscores of psychotic-like symptoms of the Neuropsychiatric Inventory (NPI), namely Delusions, Hallucination, and Agitation/Aggression.

SECONDARY OUTCOMES:
Change from Baseline in the Neuropsychiatric Inventory (NPI) total score | Baseline, Week 2, Week 10
  Neuropsychiatric Inventory (NPI), a scale that includes ten behavioral items (delusions, hallucinations, agitation, depression, anxiety, euphoria, apathy, disinhibition, irritability and aberrant motor behaviors) and two neurovegetative symptoms (sleep and appetite disorders). The evaluation was based on an interview with patients' primary caregivers. Both the frequency (/4) and the severity (/3) of each behavior were determined and a score was calculated by multiplying the frequency and the severity of each behavior observed.
Change from Baseline in the Neuropsychiatric Inventory (NPI) subscores | Baseline, Week 2, Week 10
  Neuropsychiatric Inventory (NPI) scale includes ten behavioral items (delusions, hallucinations, agitation, depression, anxiety, euphoria, apathy, disinhibition, irritability and aberrant motor behaviors) and two neurovegetative symptoms (sleep and appetite disorders). For each behavior the frequency (/4) and the severity (/3) were determined, corresponding to a subscore.
Change from Baseline in the Zarit scale score | Baseline, Week 2, Week 10
  The burden of the family caregiver was measured with the Zarit burden interview scale (completed by the caregiver). Composed of 22 questions on the physical, emotional and financial load felt. Total score /88.
Change from Baseline in the Trail Making Test (TMT) A&B performances | Baseline, Week 2, Week 10
  The TMT A&B is a task requiring a subject to connect a sequence of 25 consecutive targets on a sheet of paper, in the shortest time possible without lifting the pen from the paper. Performances are time and number of errors
Change from Baseline in the Quality of life questionnaire (Qol) | Baseline, Week 2, Week 10
  QoL was measured using the 13-item Quality of Life in Alzheimer's Disease (QOL-AD) scale (total score range 13-52; higher scores indicate better QOL). The QOL-AD scale uses a scale of 1-4 (poor, fair, good, or excellent) to rate a variety of life domains, including the patient's physical health, mood, relationships, activities, and ability to complete tasks
Change from Baseline in the Mayo Clinic fluctuations scales score | Baseline, Week 2, Week 10
  The Mayo Fluctuations Scale is a four-item questionnaire assessing the common symptoms of cognitive fluctuation shown to significantly differentiate Lewy Body Dementia from Alzheimer disease. These four items are daytime drowsiness, daytime sleepiness, disorganised thought and staring spell. Total score /4.
Change from Baseline in the percentage of errors during an "antisaccades" paradigm | Baseline, Week 2, Week 10
  Eye movements were recorded and analyzed with an eye-tracking device.
Change from Baseline in the saccades latency (in ms) during an "antisaccades" paradigm | Baseline, Week 2, Week 10
  Eye movements were recorded and analyzed with an eye-tracking device.
Change from Baseline in the mean variation of latency times (in ms) during voluntary saccades | Baseline, Week 2, Week 10
  Eye movements are recorded and analyzed with an eye-tracking device. Mean measurement is calculated from several saccades latency recorded during voluntary saccades paradigm
Change from Baseline in the frequency of square waves-jerks during horizontal eye movements paradigm | Baseline, Week 2, Week 10
  Eye movements are recorded and analyzed with an eye-tracking device. Presence, absence, frequency (number/minute) of square wave-jerks are recorded.
Change from Baseline in the frequency of fixations impairments during eye movements paradigm | Baseline, Week 2, Week 10
  Eye movements are recorded and analyzed with an eye-tracking device. Presence, absence, frequency of nystagmus, flutters or other fixations impairments
Change from Baseline in the saccades main velocity during oculomotor paradigms | Baseline, Week 2, Week 10
  This concerns saccades Main velocity (in °/sec) during vertical and horizontal paradigms. Eye movements were recorded and analyzed with an eye-tracking device.
Change from Baseline in the saccades gain during oculomotor paradigms | Baseline, Week 2, Week 10
  This concerns saccades Gain (gaze accuracy) during vertical and horizontal paradigms. Gain range 0-1. Eye movements were recorded and analyzed with an eye-tracking device.
Change from Baseline in the saccades latency during oculomotor paradigms | Baseline, Week 2, Week 10
  This concerns saccades Latency (in ms) during vertical and horizontal paradigms. Eye movements were recorded and analyzed with an eye-tracking device.

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine LOUCHART de la CHAPELLE, MD, PhD, Principal Investigator — Memory Clinic and Gerontologic center, Princess Grace Hospital (MONACO)
Locations (1):
- Clinical Research Unit-Memory Clinic / Centre de Gérontologie Clinique Rainier III / Princess Grace Hospital, Monaco, Monaco

IPD SHARING:
Plan to Share IPD: Yes
The specific individual participant data (IPD) sets to be shared would be all IPD that underlie results in a publication
Time Frame: the data will become available when summary data are published
Access Criteria: We will not share our data publicly, but we may provide it upon reasonable request to the principal investigator or the central contact person.